CLINICAL TRIAL: NCT06058520
Title: Capsule Microbiota Transplant Therapy for Hidradenitis Suppurativa
Status: Recruiting | Phase: Early Phase 1 | Type: Interventional
Sponsor: University of Minnesota (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Treatment
Other Study IDs: DERM-2023-31562
Record Dates: First submitted 2023-09-11; First posted 2023-09-28 (Actual); Last update posted 2025-12-23 (Actual); Status verified 2025-12

CONDITIONS: Hidradenitis Suppurativa
MeSH Terms: conditions — Hidradenitis Suppurativa

STUDY DESIGN:
Intervention Model Description: This study is an exploratory, randomized, double blind, placebo- controlled clinical trial. Subjects and investigators will be blinded to the Microbiota transplant therapy (MTT) and placebo arms.
Who Masked: Participant, Investigator
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: Yes | FDA-regulated Device: No

ARMS (2):
- MMT group (Experimental): patients with HS randomized to receive MTT
  Interventions: Drug: Fecal Microbiota - lyophilized
- Placebo group (Placebo Comparator): patients with HS randomized to receive placebo treatment
  Interventions: Drug: Placebo drug

INTERVENTIONS:
Drug: Fecal Microbiota - lyophilized — Patients receive 2 capsules daily for one week followed by one capsule daily for 2 weeks. MTT capsules are derived from a single donor per patient.
  Arms: MMT group
Drug: Placebo drug — The placebo consists of a mixture of trehalose and crystalline methylcellulose (Avicel) in 6:1 (w/w) ratio that is packaged in size 0 swedish orange capsules, which are then double encapsulated in size 00 natural colored capsules to make them visibly indistinguishable from encapsulated active product.
  Arms: Placebo group

SUMMARY:
HS is relatively common in the United States with a prevalence of 0.1-1.0%. 1 HS has a dramatic impact on quality of life, significantly more so than other chronic skin diseases, such as psoriasis or atopic dermatitis (AD). HS also has a large economic impact, due to frequent emergency department and inpatient care utilization, and re-hospitalization rates similar to congestive heart failure. Unfortunately, few treatment options are effective. There are currently three FDA-approved treatments for HS, including adalimumab, secukinumab, and bimekizumab, each with only 40- 60% respond to treatment and over 50% lose response within one year . The overarching goal of this pilot study is to investigate the central hypothesis that oral microbiota transplant therapy(MTT) alters the gut microbiome in patients with Hidradenitis Suppurativa (HS), influencing cutaneous microbiota via systemically absorbed gut-derived metabolites.

ELIGIBILITY:
Inclusion Criteria:

* Able and willing to provide informed consent
* English speaking
* Age >= 18years of age
* Diagnosis of hidradenitis suppurativa by a dermatologist
* Women who are not post-menopausal (at least 12 months of non-therapy induced amenorrhea) or surgically sterile (e.g. absence of ovaries and/or uterus) must remain abstinent or use a highly effective form of birth control (e.g. oral contraception, transdermal patch, barrier, intrauterine device). Periodic abstinence and early withdraw are not acceptable methods
* Able to comply to study measures in the opinion of the investigator.
* Stable doses of all medications for 30 days prior to baseline

Exclusion Criteria:

* Non-English speaking
* Refusal or inability to provide informed consent
* Planning on moving within 6 months from start of study
* Allergy to neomycin or vancomycin
* Anaphylactic food allergies
* Pregnancy, breastfeeding or planning pregnancy during study period (negative pregnancy test needed for persons of childbearing potential)
* Use of any topical or oral antibiotics within 30 days of randomization
* Use of any oral antibiotics within 90 days of randomization
* History of inflammatory bowel disease
* Extensive bowel resection (e.g., subtotal colectomy, substantial removal of small bowel)
* No major bowel surgery within 4 weeks prior to baseline or planned major surgery during the study period
* No active skin disease other than HS that could interfere with assessments

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 16 (Estimated)
Dates: Start 2023-10-01 (Actual); Primary Completion 2026-09-01 (Estimated); Study Completion 2026-09-01 (Estimated)

PRIMARY OUTCOMES:
Percent donor engraftment | Baseline, 6 weeks, 12 weeks
  Percent donor engraftment based on Bayesian, community-wide, culture-independent microbial source tracking

SECONDARY OUTCOMES:
Skin toxonomic relative abundances and diversity indices | 6 weeks, 12 weeks
  Change in skin taxonomic relative abundances and diversity indices (alpha and beta diversity) at 6 and 12 weeks compared to baseline (t- test and regression-analysis evaluating change overtime for two and three time points)
Stool toxonomic relative abundances and diversity indices | 6 weeks, 12 weeks
  Change in stool taxonomic relative abundances and diversity indices (alpha and beta diversity) at 6 and 12 weeks compared to baseline (t- test and regression-analysis evaluating change overtime for two and three time points)
Stool small chain fatty acids | 12 weeks
  Change in stool small chain fatty acids (butyrate, acetate and propionate) at 12 weeks compared to baseline
Serum small chain fatty acids | 12 weeks
  Change in serum small chain fatty acids (butyrate, acetate and propionate) at 12 weeks compared to baseline
Stool small molecule metabolites | 6 weeks, 12 weeks
  change in stool small molecule metabolites including kynurenine, tryptophan and sphingomyelins at 6 and 12 weeks compared to baseline
Physician-reported clinical response 1 | 12 weeks
  Physician-reported clinical response at 12 weeks compared to baseline measured by Hidradenitis Suppurativa Clinical Response (HiSCR)
Physician-reported clinical response 2 | 12 weeks
  Physician-reported clinical response at 12 weeks compared to baseline measured by International Hidradenitis Suppurativa Severity Score 55 (IHS4-55)
Change in IHS4 | 12 weeks
  12 weeks compared to baseline
Change in total draining tunnel count | 12 weeks
  12 weeks compared to baseline
Change in the Hidradenitis Suppurativa Activity and Severity Index | 12 weeks
  12 weeks compared to baseline
Change in Hidradenitis Suppurativa quality of life (HiSQOL) | 12 weeks
  12 weeks compared to baseline
Change in Dermatology Life Quality Index (DLQI) | 12 weeks
  12 weeks compared to baseline
Change in skin pain numerical rating scale (NRS) | 12 weeks
  12 weeks compared to baseline
Change in hidradenitis suppurativa patient global assessment | 12 weeks
  12 weeks compared to baseline

CONTACTS AND LOCATIONS:
Locations (1):
- University of Minnesota, Minneapolis, Minnesota, United States

IPD SHARING:
Plan to Share IPD: No